CLINICAL TRIAL: NCT05041062
Title: A Phase II Prospective, Open-label Trial of Perioperative Combination Nivolumab and Ipilimumab in Patients With Resectable Malignant Peritoneal Mesothelioma
Brief Title: A Study of Immunotherapy Drugs Nivolumab and Ipilimumab in Patients w/Resectable Malignant Peritoneal Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-0672
Record Dates: First submitted 2021-09-07; First posted 2021-09-10 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Mesothelioma; Peritoneal Mesothelioma
Keywords: chest cancer; abdominal cancer; lung cancer; cancer in lining of lungs
MeSH Terms: conditions — Mesothelioma; Lung Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Participants in Study Who Have Mesothelioma (Experimental): Individuals in this group will receive a combination of two immunotherapy drugs (nivolumab and ipilimumab) before and after surgery to remove their cancer. There will also be a follow up period to determine how well the drugs and surgery worked to get rid of your cancer. Your overall participation in this study (including drug treatment, surgery and follow up visits) will last for roughly one and a half years. All eligible participant who enroll in the study will participate in this group.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is an immunotherapy drug (a type of drug that helps your immune system fight cancer) that is often used with ipilimumab as the first treatment in adults with mesothelioma whose disease cannot be removed by surgery. The drug will be given as an IV infusion.
  Other Names: Opdivo; ONO-4538; BMS-936558; MDX1106
Drug: Ipilimumab — Ipilimumab is a type of immunotherapy drug known as a checkpoint inhibitor, which helps your own immune system attack cancer cells.
  Other Names: Yervoy

SUMMARY:
This study is for individuals who have peritoneal mesothelioma, a cancer of the lining of your abdominal wall and organs (the peritoneum). Doctors leading the study would like to determine the effects of treating this cancer with immunotherapy drugs (nivolumab and ipilimumab - the two study drugs that will be used in this study) before and after surgery.

Doctors hope to learn if giving these two drugs before surgery will decrease the amount of viable (live) cancer cells that remain at the time of surgery and whether it will delay the time it could take for the cancer to regrow.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of histologically or cytologically confirmed peritoneal mesothelioma, of epithelial, biphasic, or sarcomatoid subtypes
2. Have disease burden amenable to cytoreduction and hyperthermic intraperitoneal chemotherapy (HIPEC), as determined by a surgeon specializing in mesothelioma
3. Have measurable or evaluable disease based on RECIST 1.1 or on laparoscopy
4. Have no definitive evidence of visceral metastases by best staging
5. Be willing to undergo laparoscopy or mini-laparotomy for peritoneal staging
6. Adequate organ function as determined by screening labs,
7. Have an ECOG performance status of < 2
8. Be 18 years of age on day of signing informed consent
9. Be willing and able to provide written informed consent for the trial

Exclusion Criteria:

1. Is currently participating in a study of an investigational agent and received an investigational agent within 4 weeks of the first dose of treatment on this protocol
2. Has received any immunotherapy agents outside of this protocol within 4 weeks of the first dose of treatment on this protocol
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (>10 mg of prednisone daily or equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study drug.
4. Has a known history of active TB infection (Bacillus tuberculosis)
5. Has active COVID-19 infection
6. Has known history of, or any evidence of active, non-infectious pneumonitis that required steroids, or active pneumonitis
7. Has a severe hypersensitivity to nivolumab or any of its excipients
8. Has a severe hypersensitivity to ipilimumab or any of its excipients
9. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
10. Has a known additional malignancy that is progressing or required active treatment within the 3 years prior to enrollment - exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or other tumors that will not affect life expectancy
11. Has an active infection requiring systemic therapy
12. Has a known history of HIV, Hepatitis B, or Hepatitis C
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment

    1. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
    2. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.8.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
    3. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
15. Is on anticoagulation that cannot be discontinued in the perioperative period
16. Has received a live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Turaga, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants in Study Who Have Mesothelioma: Individuals in this group will receive a combination of two immunotherapy drugs (nivolumab and ipilimumab) before and after surgery to remove their cancer.
  Nivolumab: Nivolumab is an immunotherapy drug (a type of drug that helps the immune system fight cancer) that is often used with ipilimumab as the first treatment in adults with mesothelioma whose disease cannot be removed by surgery. The drug will be given as an IV infusion.
  Ipilimumab: Ipilimumab is a type of immunotherapy drug known as a checkpoint inhibitor, which helps the immune system attack cancer cells.
Period: Overall Study
Arm/Group | All Participants in Study Who Have Mesothelioma
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 54.0 [42 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Major Pathologic (Disease) Response of Tumor to Nivolumab Combined With Ipilimumab Before Surgery
Description: The response of participant's tumor to treatment with nivolumab and ipilimumab before surgery by analyzing tissue samples collected from participant during surgery for the presence of cancerous tumour cells. Major pathologic response will be defined as tissue samples containing less than or equal to 10% of residual (leftover) tumor/cancer in the tissue after surgery.
Time Frame: 24 months
Population: Data not collected.
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 0

2. Secondary Outcome: Rate of Participants Who Report Serious Side Effects to Nivolumab Combined With Ipilimumab Before Surgery (Neoadjuvant Treatment)
Description: The rate of participants who report Grade 3 or 4 serious adverse events (side effects) after taking nivolumab combined with ipilimumab before surgery. These side effects will be measured according to Common Terminology Criteria for Adverse Events v5.0 for up to 30 days after surgery.
Time Frame: 3 weeks (timeframe for surgery ) + 30 days (timeframe for assessing side effects after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Number of Participants Who Proceed to Surgery Without Delays After Receiving Nivolumab Combined With Ipilimumab
Description: Number of participants who complete treatment with nivolumab and ipilimumab before surgery and proceed to surgery without extended treatment-related delays or progression precluding surgery as assessed by clinical /study records.
Time Frame: 19 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Overall Survival of Participants Who Take Nivolumab Combined With Ipilimumab Before Surgery
Description: Overall survival of participants who receive neoadjuvant nivolumab combined with ipilimumab, defined as time from enrollment on study to death from any cause.
Time Frame: 42 Months
Population: Data not collected.
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-Free Survival of Participants Who Take Nivolumab Combined With Ipilimumab Before Surgery
Description: Progression-free survival of participants who receive neoadjuvant nivolumab combined with ipilimumab, defined as time from enrollment on study to death from any cause.
Time Frame: 42 months
Population: Data not collected.
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 0

6. Secondary Outcome: Rate of Participants Who Report Serious Side Effects to Taking Nivolumab Combined With Ipilimumab After Surgery (Adjuvant Treatment)
Description: The rate of participants who report Grade 3 or 4 serious adverse events (side effects) after taking nivolumab combined with ipilimumab after surgery. These side effects will be measured according to Common Terminology Criteria for Adverse Events v5.0.
Time Frame: 12 weeks
Population: Neither of the two enrolled patients received study drug (nivolumab/ipilimumab) after surgery.
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 0

7. Secondary Outcome: Radiologic Response to Nivolumab and Ipilimumab Before Surgery
Description: Radiologic response to nivolumab and ipilimumab before surgery using radiology images of tumor pre- and post-treatment.
Time Frame: 24 months
Population: Data not collected.
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 0

8. Secondary Outcome: Peritoneal Carcinomatosis Index (PCI) of Participants Who Taking Nivolumab Combined With Ipilimumab Before Surgery
Description: The effect of nivolumab and ipilimumab on participant's tumor as assessed by a peritoneal carcinomatosis index (PCI) score, a score determined based on the size of participant's tumor after abdominal surgery.
  The Peritoneal Cancer Index (PCI) scoring system is a diagnostic and prognostic tool. The PCI score is calculated by dividing the peritoneal (abdominal) cavity into 13 regions and assigning a score to each of the 13 regions. Each region receives a score of 0-3 based on the largest tumor size in each region. The total sum of all 13 regions is the PCI score. PCI scores can range from 0 to 39. Higher scores indicate more widespread and/or larger tumors in the peritoneal cavity.
Time Frame: 12 weeks
Population: Data not collected.
Arm/Group | All Participants in Study Who Have Mesothelioma
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | All Participants in Study Who Have Mesothelioma
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants in Study Who Have Mesothelioma (N=2)
Acute kidney injury (Renal and urinary disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants in Study Who Have Mesothelioma (N=2)
Pain (General disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Respiratory, thoracic and mediastinal disorders-Other (Respiratory, thoracic and mediastinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Rash (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT05041062/Prot_SAP_000.pdf